CLINICAL TRIAL: NCT03052816
Title: ICE-T Postoperative Multimodal Pain Regimen Compared to the Standard Regimen in Same Day Vaginal Pelvic Reconstructive Surgery: a Randomized Controlled Trial
Brief Title: Ice T Postoperative Multimodal Pain Regimen in FPMRS Surgery
Acronym: ICET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00498
Record Dates: First submitted 2017-01-31; First posted 2017-02-14 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative; Pelvic Organ Prolapse
MeSH Terms: conditions — Pain, Postoperative; Pelvic Organ Prolapse | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ICE T (Experimental): 1. ICE PACKS applied to the perineum every hour for 20 minutes ATC until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV Q3 hr PRN for breakthrough pain.
  5. Patients will be discharged home with PO Tylenol and PO toradol PRN.
  Interventions: Drug: Ice T
- Standard (Active Comparator): 1. Motrin 600mg PO Q4h PRN pain 1-3
  2. Percocet 1 tab PO Q4-6 hours PRN 4-6 pain
  3. Percocet 2 tabs PO Q 7-10 hours PRN 7-10 pain
  4. Patients will receive dilaudid 0.2mg IV Q3 hr PRN for breakthrough pain.
  5. Patients will be discharged home with Motrin and Percocet for pain PRN.
  Interventions: Drug: Motrin/Percocet/Dilaudid for breakthrough

INTERVENTIONS:
Drug: Ice T — Ice/Tylenol/Toradol with dilaudid for breakthrough
  Arms: ICE T
Drug: Motrin/Percocet/Dilaudid for breakthrough — Standard regimen
  Arms: Standard

SUMMARY:
The purpose of this randomized controlled trial is to determine whether, "ICE-T," a novel multimodal postoperative pain regimen composed of around the clock ice packs, toradol, and tylenol, has improved pain control intake compared to the standard postoperative pain regimen in patients undergoing vaginal pelvic floor reconstructive surgery.

DETAILED DESCRIPTION:
Pelvic floor disorders involve a myriad of complicated, interwoven clinical conditions that involve pelvic organ prolapse, urinary incontinence, fecal incontinence, and other pathology involving the genital and lower urinary tract. It is estimated that pelvic floor disorders affect up to 25% of all adult women in the United States with increasing prevalence with age. By the age of sixty, 1 in 9 women will undergo surgical intervention for pelvic organ prolapse and/or incontinence, increasing to 1 in 5 by the age of 80. As the population in the United States ages, the demand for healthcare for pelvic floor disorders is estimated to increase up to 40% in the next 30 years.

Despite the prevalence of surgery performed for pelvic floor disorders, there is a paucity of data on postoperative pain control that is dedicated to female pelvic reconstructive surgery. In a recent review, there was only one study that evaluated postoperative pain control after vaginal reconstructive surgery, and the mainstay of therapy was opioid driven. Generally, postoperative pain control in gynecologic surgery has been opioid driven, frequently involving multiple narcotics for analgesia, resulting opioid related complications, including nausea, vomiting, constipation, urinary retention, and central nervous system side effects In an effort to combat opioid use in gynecologic and female pelvic reconstructive surgery, multimodal therapy has been gaining momentum with goals of improved pain control and decreased opioid requirements. Ice packs, toradol, and acetaminophen have been used in various trials to decrease postoperative opioid requirements in various surgeries.

Ice packs have been shown to be effective in the treatment of postoperative pain after abdominal midline incisions. A Cochrane Review of patients subject to post vaginal delivery perineal cooling included 10 randomized controlled trials with1825 patients with some evidence that local cooling in the form of ice packs, cold gel packs, cold/ice backs may be effective in pain relief.

Toradol has been extensively studied in a multitude of surgeries including spinal, obstetric, orthopedic, urologic, and gynecologic. It has been administered preemptively, intraoperatively, and postoperatively for pain control with evidence that toradol decreases postoperative subjective pain scores and decreased narcotic use.

Acetaminophen is mainstay for postoperative pain control as part of multimodal pain regimens to complement other, opioid sparing medications in a multitude of surgeries including abdominal hysterectomy.

Therefore, the purpose of this randomized controlled study is to determine whether, "ICE-T" a novel multimodal postoperative pain regimen composed of around the clock ice packs, toradol, and tylenol, has improved pain control and decrease opioid intake compared to the standard postoperative pain regimen in patients undergoing vaginal pelvic floor reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are the following:
* Consenting, English speaking women between ages 18 and 80 who will undergo same day vaginal female pelvic reconstructive surgery at MetroHealth Medical Center
* Ability to read VAS Scores
* Specific vaginal procedures include, but are not limited to:

  * Periurethral bulking
  * Perineoplasty
  * Complete vaginectomy
  * Le Forte colpocleisis
  * Anterior repair
  * Posterior repair
  * Enterocele repair
  * Anterior and posterior repair
  * Anterior, posterior and enterocele repair
  * Transvaginal mesh use
  * Sacrospinous ligament fixation
  * Uterosacral ligament suspension
  * Vaginal paravaginal defect repair
  * Midurethral Sling
  * Sphincteroplasty
  * Vaginal hysterectomy, for uterus 250 g or less
  * Vaginal hysterectomy, for uterus 250 g or less; with removal of tube(s), and/or ovary(s)
  * Vaginal hysterectomy, for uterus 250 g or less; with removal of tube(s), and/or ovary(s), with repair of enterocele
  * Vaginal hysterectomy, for uterus 250 g or less; with repair of enterocele
  * Vaginal hysterectomy, for uterus greater than 250 g
  * Vaginal hysterectomy, for uterus greater than 250 g; with removal of tube(s) and/or ovary(s)
  * Vaginal hysterectomy, for uterus greater than 250 g; with removal of tube(s) and/or ovary(s), with repair of enterocele
  * Vaginal hysterectomy, for uterus greater than 250 g; with repair of enterocele

Exclusion Criteria:

* The exclusion criteria are the following:
* History of chronic pelvic pain
* Abdominal surgery
* Laparoscopic surgery
* History of psychiatric disease
* Currently taking analgesic medications
* Currently taking sedatives
* Liver disease
* Renal disease with CrCl < 60cc/min.
* History of burns from application of ice.
* Women who did not consent for the study.
* Intraoperative concern for increased blood loss
* Unable to speak English
* Unable to understand VAS Scores
* Undergoing concomitant abdominal or laparoscopic procedures.
* Allergy to motrin, toradol, Percocet, Tylenol
* Active or history of peptic ulcer disease
* History of GI bleeding or perforation
* Hemorrhagic diathesis
* Severe uncontrolled heart failure
* Inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients who undergo same day (<24 hour) female pelvic reconstructive surgery
Enrollment: 66 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrikovets A, Sheyn D, Sun HH, Chapman GC, Mahajan ST, Pollard RR, El-Nashar SA, Hijaz AK, Mangel J. Multimodal opioid-sparing postoperative pain regimen compared with the standard postoperative pain regimen in vaginal pelvic reconstructive surgery: a multicenter randomized controlled trial. Am J Obstet Gynecol. 2019 Nov;221(5):511.e1-511.e10. doi: 10.1016/j.ajog.2019.06.002. Epub 2019 Jun 12. PMID 31201808

FDAAA 801 VIOLATIONS:
- Correction Confirmed — The responsible party has corrected the violation. — issued 2021-12-20, released 2021-10-03, posted 2022-01-06
- Violation Identified — Failure to Submit. The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2021-08-31, released 2018-12-15, posted 2021-09-03

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study approved January 30th, 2017. First patient recruited April 2017. Between April 2017 and April 2018, 138 women who were scheduled for surgery were assessed. 72 patients were excluded. Sixty-six patients were randomized to the ICE-T or Standard protocols. Of the 33 patients who were randomized to the ICE-T regimen, three were excluded after randomization. Ultimately, thirty patients in the ICE-T arm and 33 patients in the Standard arm were analyzed.
Pre-assignment Details: 138 Patients assessed for eligibility. 72 patients excluded: 55 not meeting inclusion criteria and 17 declined to participate.
  66 were randomized.
Groups:
- ICE T Postoperative Pain Regimen: 1. ICE PACKS applied to the perineum every hour for 20 minutes ATC until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV Q3 hr PRN for breakthrough pain.
  5. Patients will be discharged home with PO Tylenol and PO toradol PRN.
  Ice T: Ice/Tylenol/Toradol with dilaudid for breakthrough
- Standard Postoperative Pain Regimen: 1. Motrin 600mg PO Q4h PRN pain 1-3
  2. Percocet 1 tab PO Q4-6 hours PRN 4-6 pain
  3. Percocet 2 tabs PO Q 7-10 hours PRN 7-10 pain
  4. Patients will receive dilaudid 0.2mg IV Q3 hr PRN for breakthrough pain.
  5. Patients will be discharged home with Motrin and Percocet for pain PRN.
  Motrin/Percocet/Dilaudid for breakthrough: Standard regimen
Period: Overall Study
Arm/Group | ICE T Postoperative Pain Regimen | Standard Postoperative Pain Regimen
Started | 33 | 33
Completed | 30 | 33
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Desired opioids | 2 | 0

BASELINE CHARACTERISTICS:
Population: There were 66 total patients that were randomized. 3 patients were excluded from the ICE-T arm whereas non were excluded from the Standard arm. 30 patients analyzed in the ICE-T arm and 33 patients in the Standard arm.
Groups:
- ICE T: • At the end of surgery patients receive 30mg of IV ketorolac.
  Once out of PACU patients receive:
  * ICE PACKS applied to the perineum Q2h for 20 minutes ATC until discharge
  * Ketorolac 30mg IV Q6h ATC until discharge
  * Acetaminophen 1g PO Q6h ATC until discharge
  * Hydromorphone 0.2mg IV Q3h PRN for breakthrough pain
  * Patients are discharged home with:
    1. Acetaminophen 1 gram PO every 6 hours PRN pain 1-5 #60
    2. Ketorolac 10mg PO every 6 hours PRN pain #6-10 #16
- STANDARD: • At the end of surgery patients receive 30mg of IV ketorolac.
  Once out of PACU patients receive:
  * Ibuprofen 600mg PO Q4h PRN pain 1-3
  * Acetaminophen/oxycodone 5mg/325mg 1 tablet PO Q4-6h PRN pain 4-6
  * Acetaminophen/oxycodone 5mg/325mg 2 tablets PO Q4-6h PRN pain 7-10
  * Hydromorphone 0.2mg IV Q3h PRN for breakthrough pain
  * Patients are discharged home with:
    1. Ibuprofen 600mg PO Q8h PRN pain 1-5 #60
    2. Acetaminophen/oxycodone 5mg/325mg 1-2 tablets Q4-6h PRN pain 6-10 #16
- Total: Total of all reporting groups
Arm/Group | ICE T | STANDARD | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.1) | 59.8 (12.7) | 60.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 20 | 28 | 48
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scores (VAS)
Description: Visual Analog Scores (VAS) Scores in the morning of post op day 1. The VAS is a 100mm scale with a score of no pain on the left of the scale, indicating a score of 0, and a score of worst pain on the right, indicating a score of 10. Patient is instructed to score the scale where they feel is appropriate. Each demarcation in between marks is 10mm and after the patient marks their score it is measured using mm from 0mm-100mm. A score of 0 is 0mm and a score of 10 is 100mm.
Time Frame: Visual Analog Scores (VAS) Score in the morning of post op day 1 at 7am.
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- ICE T: 1. ICE PACKS applied to the perineum every hour for 20 minutes ATC until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV Q3 hr PRN for breakthrough pain.
  5. Patients will be discharged home with PO Tylenol and PO toradol PRN.
  Ice T: Ice/Tylenol/Toradol with dilaudid for breakthrough
- Standard: 1. Motrin 600mg PO Q4h PRN pain 1-3
  2. Percocet 1 tab PO Q4-6 hours PRN 4-6 pain
  3. Percocet 2 tabs PO Q 7-10 hours PRN 7-10 pain
  4. Patients will receive dilaudid 0.2mg IV Q3 hr PRN for breakthrough pain.
  5. Patients will be discharged home with Motrin and Percocet for pain PRN.
  Motrin/Percocet/Dilaudid for breakthrough: Standard regimen
Arm/Group | ICE T | Standard
Number analyzed (Participants) | 30 | 33
mm | 20 [10 to 20] | 40 [20 to 50]

2. Secondary Outcome: VAS Scores at 4 Hours Post Surgery
Description: VAS Scores at 4 hours post surgery. The VAS is a 100mm scale with a score of no pain on the left of the scale, indicating a score of 0, and a score of worst pain on the right, indicating a score of 10. Patient is instructed to score the scale where they feel is appropriate. Each demarcation in between marks is 10mm and after the patient marks their score it is measured using mm from 0mm-100mm. A score of 0 is 0mm and a score of 10 is 100mm.
Time Frame: VAS Scores at 4 hours post surgery
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | ICE T | Standard
Number analyzed (Participants) | 30 | 33
mm | 35 [0 to 70] | 50 [30 to 80]

3. Secondary Outcome: VAS Scores 96 Hours After Surgery
Description: VAS Scores 96 hours after surgery. The VAS is a 100mm scale with a score of no pain on the left of the scale, indicating a score of 0, and a score of worst pain on the right, indicating a score of 10. Patient is instructed to score the scale where they feel is appropriate. Each demarcation in between marks is 10mm and after the patient marks their score it is measured using mm from 0mm-100mm. A score of 0 is 0mm and a score of 10 is 100mm.
Time Frame: VAS Scores 96 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
mm | 20 [0 to 30] | 30 [15 to 50]

4. Secondary Outcome: Quality of Recovery Scores on Post op Day 1
Description: Quality of Recovery scores on post op day 1. The QoR-40 is a 40-item quality of recovery score measuring 5 dimensions: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item is rated on a 5-point Likert scale. The QoR-40 has a possible score of 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). It was specifically designed to measure a patient's health status after surgery and anesthesia, and it has been proposed as a measure of outcome in clinical trials.
Time Frame: Quality of Recovery scores on post op day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
score on a scale | 182 [158 to 189] | 173 [164 to 182]

5. Secondary Outcome: Satisfaction Scores in the Morning After Surgery (7AM)
Description: Satisfaction scores in the morning after surgery (7AM). The satisfaction score is a numerical score from 0-10 with a score of 0 indicating very dissatisfied on the left of the scale and 10 indicating very satisfied on the right of the scale.
Time Frame: Satisfaction scores in the morning after surgery (7AM)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
score on a scale | 10 [8 to 10] | 10 [8 to 10]

6. Secondary Outcome: Satisfaction Scores 96 Hours After Surgery
Description: Satisfaction scores 96 hours after surgery. The satisfaction score is a numerical score from 0-10 with a score of 0 indicating very dissatisfied on the left of the scale and 10 indicating very satisfied on the right of the scale.
Time Frame: Satisfaction scores 96 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
score on a scale | 10 [8.5 to 10] | 9 [8 to 10]

7. Secondary Outcome: Length of Stay
Description: Length of time from the end of surgery to discharge home from the hospital, assessed up to 1 week.
Time Frame: Time from end of surgery to discharge home from hospital, assessed up to 1 week.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
hours | 24.1 (3.1) | 24.1 (5.4)

8. Secondary Outcome: Total Dose of Opioids Administered During Hospitalization
Description: Total dose of opioids administered during hospitalization in morphine equivalents upon hospital discharge.
Time Frame: Total dose of opioids administered during hospitalization in morphine equivalents from the end of surgery to discharge up to 1 week
Measure: Mean (Standard Deviation); unit: milligrams of oral morphine equivalents
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
milligrams of oral morphine equivalents | 55.7 (31.2) | 91.2 (38.9)

9. Secondary Outcome: Postoperative Nausea and Vomiting at 7AM After Surgery
Description: Number of patients with postoperative nausea and vomiting at 7AM after surgery
Time Frame: Postoperative nausea and vomiting from the time to end of surgery until 7AM after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
Participants | 14 | 18

10. Secondary Outcome: Number of Participants With Urinary Retention.
Description: Number of participants with urinary retention (discharge home with foley)
Time Frame: Number of participants with urinary retention (discharge home with foley) measured on day patient is discharged home/study completion up to 1 week.
Measure: Count of Participants; unit: Participants
Arm/Group | ICE T | STANDARD
Number analyzed (Participants) | 30 | 33
Participants | 5 | 7

ADVERSE EVENTS:
Time Frame: Each patient was assessed for adverse events during the course of the entire study extending one month after completion of recruitment to allow for one month after surgery for each patient recruited.
Description: An independent data and safety monitoring physician in the Department of Obstetrics and Gynecology at both institutions oversaw the progress of the study.
Arm/Group | ICE T | Standard
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT03052816/Prot_SAP_002.pdf